CLINICAL TRIAL: NCT06436196
Title: Video Laryngoscopy Versus Direct Laryngoscopy for Elective Airway Management in Pediatrics Anesthesia, Comparison of Out-comes
Brief Title: Video Laryngoscopy vs Direct Laryngoscopy in Paediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Muhammad Ilyas, Assistant Professor, Watim Medical & Dental College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CMH/614
Record Dates: First submitted 2024-05-19; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Endotracheal Tube Wrongly Placed During Anesthetic Procedure

STUDY DESIGN:
Intervention Model Description: Comparitive study between 2 groups.
Who Masked: Participant
Masking Description: Participants are not aware of the method which will be used to secure their airway.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Laryngoscopy Group (Active Comparator): Group of patients in which standard direct laryngoscopy will be used to secure airway.
  Interventions: Device: Direct laryngoscope
- Video Laryngoscopy group (Active Comparator): Group of patients in which Video Laryngoscopy will be used to secure airways.
  Interventions: Device: Video Laryngoscope

INTERVENTIONS:
Device: Video Laryngoscope — Use of Video laryngoscope to secure airway
  Arms: Video Laryngoscopy group
Device: Direct laryngoscope — Macintosh or Miller's laryngoscopes used to secure paediatric airways
  Arms: Direct Laryngoscopy Group

SUMMARY:
The goal of this interventional study is to compare the effectiveness of direct laryngoscopy vs. video laryngoscopy in paediatric population aged 2 to 8 years presenting for elective surgeries having uncomplicated airways.

The primary outcome measures include:

1. Time taken for succesful insertion and confirmation of ETT in patients using both techniques seprately.
2. Rate of complications and failed attempts compared between both modalities.

DETAILED DESCRIPTION:
The comparision of efficacy of Video Laryngoscopy for pediatric airway vs Direct Laryngoscopy is the goal of this study, Safety of the patients will be the utmost priority with careful case selection alongwith proper informed detailed consent from the guardians of the children.

PROCEDURE:

After induction of General Anesthesia four minutes of proper bag mask ventilation to allow for proper intubating conditions will be done. The time taken from the insertion of the laryngoscopic blade to the best glottic view acheived by the specific technique will be noted seperately and then the time to the succesful acheivement of lung inflation with the proper placement of ETT will be noted seperately, both of these parameters will be recorded.

If in a patient airway is not secured even after 3 attempts by a specific technique the technique would be altered and patient would be excluded from our research.

MATERIALS:

Randomized allotment of patients into the 2 groups i.e Direct Laryngoscopy and Video Laryngoscopy would be done.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients of age between 2 - 8 years,
* American Society of Anesthesiologist (ASA) grades I-II Children
* Cormack-Lehane grade I, II and III who will need airway management for elective surgery under general anesthesia.

Exclusion Criteria:

* Patients with abnormal airway anatomy,
* Obese patients,
* Emergency surgery,
* Congenital syndrome involving any major organs
* Patients' guardians unwilling to participate .
* Patients in whom airway is not secured with a specific technique even after three attempts.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
.Time taken to acheive the best possible view of the glottis. | 4 Min. post muscle relaxant administration to 6 Min. post muscle relaxant administration
  The time from insertion of laryngoscope in the mouth to the best possible view of the glottis.
Time taken to acheive succesful Endotracheal Intubation. | 4 Min 30 seconds post muscle relaxant administration to 7 Min post muscel relaxant administration.
  The time from the insertion of the laryngoscopic blade in the mouth to the correct placement of ETT confirmed by the waveform capnorgraphy.
No. of Intubation attempts needed | 4 Min. post muscle relaxation administration to 15 Min. post muscle relaxant administration.
  Total No. of attempts(max 3 attempts with the same technique) to secure airway.

SECONDARY OUTCOMES:
Hemodynamic changes at different intervals. | During attempts to 1 min, 5 min, and 10 min post succesful intubation.
  Changes in heart rate will be assesed during attempts and to a fixed amount of time after succesfully securing the airways.
Hemodynamic changes at different intervals. | During attempts to 1 min, 5 min, and 10 min post succesful intubation.
  Changes in blood pressure will be assesed during attempts and to a fixed amount of time after succesfully securing the airways.

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Millitary Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The outcomes of the study will be shared eventually once concluded
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Undecided
Access Criteria: not yet Decided

REFERENCES:
- [Background] Rabiner JE, Auerbach M, Avner JR, Daswani D, Khine H. Comparison of GlideScope Videolaryngoscopy to Direct Laryngoscopy for Intubation of a Pediatric Simulator by Novice Physicians. Emerg Med Int. 2013;2013:407547. doi: 10.1155/2013/407547. Epub 2013 Oct 31. PMID 24288617
- [Background] Sinha R, Sharma A, Ray BR, Kumar Pandey R, Darlong V, Punj J, Chandralekha C, Upadhyay AD. Comparison of the Success of Two Techniques for the Endotracheal Intubation with C-MAC Video Laryngoscope Miller Blade in Children: A Prospective Randomized Study. Anesthesiol Res Pract. 2016;2016:4196813. doi: 10.1155/2016/4196813. Epub 2016 May 15. PMID 27293429
- [Background] Myatra SN, Patwa A, Divatia JV. Videolaryngoscopy for all intubations: Is direct laryngoscopy obsolete? Indian J Anaesth. 2022 Mar;66(3):169-173. doi: 10.4103/ija.ija_234_22. Epub 2022 Mar 24. No abstract available. PMID 35497693
- [Background] Zhou M, Xi X, Li M, Wang S, Liu Z, Liu JQ. Video Laryngoscopy Improves the Success of Neonatal Tracheal Intubation for Novices but Not for Experienced Medical Staff. Front Pediatr. 2020 Aug 6;8:445. doi: 10.3389/fped.2020.00445. eCollection 2020. PMID 32850555